CLINICAL TRIAL: NCT01609777
Title: HandSAFE - Development and Evaluation of a Handover Tool for Doctors and Nurses
Acronym: HandSAFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HandSAFE
Record Dates: First submitted 2012-04-11; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Complications of Medical Care, Nec in ICD9CM_2011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Handover with SBAR (Other): Handover with handover tool.
  Interventions: Procedure: SBAR

INTERVENTIONS:
Procedure: SBAR — situation, background, assessment, recommendation

SUMMARY:
A handover Tool for doctors and nurses improves the quality of handovers compared to handovers that are being conducted without a tool.

In the present study the investigators will develop and evaluate a handover Tool for doctors and nurses. The investigators seek to answer the following research questions:

1. Does the tool improve quality (i.e. efficiency and accuracy)?
2. Does the tool improve safety relevant attitude an perceived team collaboration?

DETAILED DESCRIPTION:
Medical transfers in the ICU are a critical part of patient care. Ensuring consistency of information that is passed on within the intensive care unit i.e. from shift to shift or between different functional areas (eg ICU to surgery) is ensured. Incorrect, incomplete or incomprehensible information in this context can have severe consequences and jeopardize patient safety. Research on handovers from other high risk organizations that are associated with a high risk of error, such as space flight control centers has shown potential consequences that result from incomplete handovers. Apart from a flawed mental model about the state of the system, the respective recipient of the handover are not able to anticipate possible future events and respond accordingly. The main barriers to implement effective handover in the medical setting are the following factors: The medical and clinical context (constant background noise and lack of privacy); the organizational hierarchy and status differences, which may lead the submitter to stress, as well as linguistic and cultural barriers that may impede further communication.

To counter these barriers, a variety of memory aids (tools) have been designed to structure the handover along defined cornerstones. Examples of such handover tools are LAURS(Listen, Accept, Utilize, Reframe, Suggest) and SBAR (Situation, Background, Assessment, Recommendation). These memory aids facilitate a problem-centered and consistent delivery of information.

This however neglect a crucial fact: from a psychological perspective, the intensive care unit presents a multi-team system. This means that different functional groups (Senior doctors, assistant doctors and nurses) work together towards a common goal, ie the treatment of a patient. However handovers occur mostly parallel with different functional areas, which hampers the consistent exchange of information between the groups. This in turn may reduce team effectiveness and lead to errors in the treatment of a patient.

For this reason, a handover tool not only supports the information flow within a function group, but also between the various functional groups. The previous research on communication between physicians and nurses suggests that the perceived psychological safety is an important prerequisite for overcoming the perceived status differences, and thus for effective and efficient teamwork. Another crucial variable for the joint achievement of a goal is the degree of perceived team collaboration i.e. cooperation between doctors and nurses. If these two parameters - psychological safety and team collaboration - are not met or are insufficient, this may lead not only to lack of information, but also to reactance against the other group. This in turn can lead to inefficient or faulty handovers and thus fatally compromise patient safety.

The aim of the proposed study, therefore, is the development and evaluation is a tool - handSAFE - designed to increase the problem-centered structure of handovers.

ELIGIBILITY:
Inclusion criteria:

* Inclusion criteria are: doctors and nurses with a minimum of 12 moths of work experience.

Exclusion criteria:

* Exclusion criteria: staff members that deny participation or don't meet the inclusion criteria

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Measurement time 4: training of the newly developed handover Tool in the patient simulator | 6 months
  Outcome measured by video-assisted analysis of the handovers and questionnaires pre- and post interventional.
Duration of handovers | 6 Month
  Measurement of the handover duration before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Bastian Grande, MD, Principal Investigator — University Hospital Zurich, Institute of Anaesthesiology
Locations (1):
- University Hospital Zurich, Institute of Anaesthesiology, Zurich, Canton of Zurich, Switzerland